CLINICAL TRIAL: NCT03542526
Title: Relationship of Different Electrocardiographic Parameters and Ambulatory Blood Pressure Parameters to Detect Left Ventricular Hypertrophy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Sadeq, cardiology resident, principle investigator, Assiut University
Other Study IDs: LVHTN
Record Dates: First submitted 2018-03-27; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: electrogradiogram — 12 lead ecg ambulatory blood prussre
  Other Names: blood measuring device
Device: ambulatory blood prussre — ambulatory blood pressure to measure blood pressure

SUMMARY:
To review the accuracy of electrocardiography in screening for left ventricular hypertrophy in patients with hypertension.

DETAILED DESCRIPTION:
Arterial hypertension is a major cause of coronary heart disease, stroke, and heart failure. Several studies have shown that left ventricular hypertrophy is an important risk factor in patients with hypertension, leading to a fivefold to 10-fold increase in cardiovascular risk,1 2 3 4 5 which is similar to the increase seen in patients with a history of myocardial infarction.6 The presence of left ventricular hypertrophy, in addition to hypertension, thus has important implications for assessing risk and managing patients, including decisions on interventions other than antihypertensive treatment, such as lipid lowering treatment and lifestyle modifications.7 8 Accurate and early diagnosis of left ventricular hypertrophy is therefore an important component of the care of patients with hypertension.

Decisions about treatment should be based on assessments of hypertensive target organ damage and overall cardiovascular risk. The appropriate diagnostic work-up of suspected left ventricular hypertrophy in patients with hypertension is less clear, however. There is many electrocardiographic indexes for the diagnosis of left ventricular hypertrophy, based on the standard 12 lead electrocardiogram, have been described. Many of the proposed indexes have remained anecdotal, but others are commonly used, including the Sokolow-Lyon index,9 the Cornell voltage index,10 the Cornell product index,11 the Gubner index,12 and the Romhilt-Estes scores.13 However, debate about their comparative diagnostic value continues.14 15 We did a systematic review to clarify the accuracy of different electrocardiographic indexes, with emphasis on their ability to rule out left ventricular hypertrophy in patients with arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

Patients ranging from 20t o 80 years attending the hypertension outpatient clinic for ambulatory blood pressure measurement will be consecutively enrolled

Exclusion Criteria:

1. Patients with ischemic heart disease.
2. Patients with advanced respiratory, renal, or hepatic disease
3. Patients with uninterpretable ECG or ABPM recordings

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients attending the Hypertension outpatient clinic over two year duration starting from November 2018, will be consecutively enrolled
Sampling Method: Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
minimize complicate of hypertension | 1 years
  screening with hypertensive patient

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
to maintain the privacy of the protocol

REFERENCES:
- [Background] Jain A, Tandri H, Dalal D, Chahal H, Soliman EZ, Prineas RJ, Folsom AR, Lima JA, Bluemke DA. Diagnostic and prognostic utility of electrocardiography for left ventricular hypertrophy defined by magnetic resonance imaging in relationship to ethnicity: the Multi-Ethnic Study of Atherosclerosis (MESA). Am Heart J. 2010 Apr;159(4):652-8. doi: 10.1016/j.ahj.2009.12.035. PMID 20362725
- [Background] Pewsner D, Juni P, Egger M, Battaglia M, Sundstrom J, Bachmann LM. Accuracy of electrocardiography in diagnosis of left ventricular hypertrophy in arterial hypertension: systematic review. BMJ. 2007 Oct 6;335(7622):711. doi: 10.1136/bmj.39276.636354.AE. Epub 2007 Aug 28. PMID 17726091
- See also: Diagnostic and Prognostic Utility of ECG for Left Ventricular Hypertrophy Defined by MRI in Relationship to Ethnicity: The Multi-Ethnic Study of Atherosclerosis (MESA) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2856691/
- See also: Accuracy of electrocardiography in diagnosis of left ventricular hypertrophy in arterial hypertension: systematic review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2001078/
- See also: Ambulatory blood pressure — https://en.wikipedia.org/wiki/Ambulatory_blood_pressure